CLINICAL TRIAL: NCT02190383
Title: Within Subject Design on the Efficacy of Habit Reversal Treatment Programme in Children and Adolescents With Tics
Brief Title: Efficacy of a Habit Reversal Treatment on Tic-symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Manfred Doepfner, Leading psychologist at the Department of Childhood and Adolescence Psychiatry, University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THICS-Study 2
Record Dates: First submitted 2014-04-14; First posted 2014-07-15 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Tic-Disorder
Keywords: Tic-Disorder, Tourette-Disorder, Habit Reversal Training
MeSH Terms: conditions — Tics; Tourette Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Habit Reversal Training (Experimental): At first patients get informed about Tics in general. Then the individual Tics are specified and the tic-reaction is looked at further. The Tic-Symptoms are observed and the premonitory urge is specified. For all individual tics a specific reversal movement is developed. Relaxation methods are introduced.
  Interventions: Behavioral: Habit Reversal Training

INTERVENTIONS:
Behavioral: Habit Reversal Training — awareness training, competing response training

SUMMARY:
The main purpose of this study is to evaluate the efficacy of a habit reversal based treatment programme in children and adolescents aged 8 to 18 years with tic disorders.

DETAILED DESCRIPTION:
The main purpose of this study is to evaluate the efficacy of a habit reversal based treatment programme for children and adolescents with tic disorders. This habit reversal treatment programme was developed at the Department of Child and Adolescent Psychiatry and Psychotherapy at the University of Cologne and has already been evaluated in a pilot-study (Woitecki & Döpfner, 2011, 2012).

ELIGIBILITY:
Inclusion Criteria:

* 8-18 years
* Diagnosis of chronic motor or vocal Tic (F95.1) or Tourette-Syndrome (F95.2)
* YGTSS total score F95.2>13, F95.1>9
* Tics are the main problems
* IQ>80
* If medication, then has been stable for at least one months in medicated patients
* No change in medication treatment is planned
* Ability to participate in weekly outpatient treatment
* Acceptance of randomization

Exclusion Criteria:

* Diagnosis of Autism Spectrum Disorder or Psychosis
* Parallel continuous psychotherapy of tics or comorbid

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Change in Symptom Checklist for Tic-Symptoms (FBB-TIC), parent rating | Baseline (T0), after 8 weeks (T1), 16 weeks (T2) and 24weeks (T3)
  The FBB-TIC is used to assess Tic-Symptoms according to DSM-IV and ICD-10 rated by parents

SECONDARY OUTCOMES:
Change in Symptom Checklist for Tic-Symptoms (FBB-/SBB-TIC), Teacher-/self-rating | Baseline (T0), after 8 weeks (T1), 16 weeks (T2) and 24weeks (T3)
  The SBB-TIC is used to assess Tic-Symptoms according to DSM-IV and ICD-10 rated by parents
Change in Symptom Checklist for Tic-Symptoms, clinical rating | Baseline (T0), after 8 weeks (T1), 16 weeks (T2) and 24 weeks (T3)
  The Checklist is used to assess Tic-Symptoms according to DSM-IV and ICD-10 rated by clinicians
Change of comorbid ADHD Symptoms (FBB/SBB-ADHD), parent, teacher and self-rating | T0, after 8 weeks (T1), 24weeks (T3)
  The Symptom Checklist for Attention Deficit/Hyperactivity Disorder (FBB-/SBB-ADHS) assess all symptom criteria according to DSM IV and ICD-10.
Change of comorbid OCD Symptoms (ZWIK-E), parent-rating | T0, after 8 weeks (T1), 24 weeks (T3)
  The ZWIK assess OCD criteria.
Change of comorbid Symptoms (CBCL/TRF/YSR), parent-/teacher-/self-rating | T0, after 8weeks (T1), 24weeks (T3)
  The CBCL, TRF and YSR assess a variation of different criteria.
Change in Tic-Symptoms (YGTSS-TIC), overall score | Baseline (T0), after 8 weeks (T1), 16 weeks (T2) and 24weeks (T3)
  The YGTSS is used to assess Tic-Symptoms in a semi structured interview with parents and patients
Change in Tic-Symptoms (observation) | Between T1 and T3 up to 16 weeks, during each session/week
  Tic symptoms are observed through video tapes and are rated through clinicians.
Change in self-esteem (Harter-Scale-SBB)(self rating) | T0, after 8 weeks (T1), 24weeks (T3)
  The Harter-Scale is used to assess self-esteem

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Döpfner, Prof. Dr., Study Director — Department of Childhood and Adolescent Psychiatry and Psychotherapy
Locations (1):
- University Hospital of Cologne, Department of Childhood and Adolescent Psychiatry and Psychotherapy, Cologne, Germany

REFERENCES:
- [Background] Woitecki K, Dopfner M. [Changes in comorbid symptoms and subjective interference in a habit reversal therapy in children with chronic tic disorder - a pilot study]. Z Kinder Jugendpsychiatr Psychother. 2012 May;40(3):181-90. doi: 10.1024/1422-4917/a000168. German. PMID 22532110
- [Background] Woitecki K, Dopfner M. [Effects of habit reversal training in children with chronic tic disorder - a pilot study]. Z Kinder Jugendpsychiatr Psychother. 2011 Nov;39(6):387-97. doi: 10.1024/1422-4917/a000137. German. PMID 22031011
- [Background] Woitecki, K. & Döpfner, M. (2014). Therapieprogramm für Kinder und Jugendliche mit Tic-Störungen (THICS). Göttingen: Hogrefe.